CLINICAL TRIAL: NCT04844476
Title: Relationship Between Fear of Falling and Balance, Posture, Spasticity and Functional Independence in Chronic Stroke Patients
Brief Title: Fear of Fall Related Factors in Chronic Stroke
Status: Completed | Type: Observational
Sponsor: Izmir Katip Celebi University (Other)
Responsible Party: Principal Investigator, Nese Olmez Sarikaya, Professor Doctor, Izmir Katip Celebi University
Other Study IDs: Fearoffallstroke
Record Dates: First submitted 2021-04-13; First posted 2021-04-14 (Actual); Last update posted 2022-04-05 (Actual); Status verified 2022-04

CONDITIONS: Stroke; Fall
Keywords: Stroke; hemiplegia; falls; fear; posture
MeSH Terms: conditions — Stroke; Hemiplegia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Some stroke survivors develop a fear of falling(FoF) which may exist with or without a prior fall. Fear of fall can be defined as decreased perceived self efficacy or confidence in maintaining balance while completing regular activities. FoF may impair rehabilitation and recovery. Determination of FoF related factors will help to identify interventions needed to decrease FoF. Mostly fear of fall related factors have been studied in acute stroke patients, limited data are available for patients with chronic stroke. The objective of this study is to evaluate frequency of FoF in chronic(>6 months) stroke patients and investigate relationship between FoF and balance, posture,spasticity and activities of daily living. The Turkish Version of the Modified Falls Efficacy Scale was used to measure FoF. Also a single-item dichotomous question "Are you afraid of falling? (Yes/No)" will be asked.

DETAILED DESCRIPTION:
In this observational study, chronic(>6 months) stroke patients who admitted to Physical Medicine and Rehabilitation outpatient clinic, older than 50 years old will be included. Sociodemographic and medical data including patients' age, gender, height, weight, body mass index, contact information, marital status, educational status, plegia side, stroke etiology, time after stroke, accompanying diseases, medications used, fear of falling (yes/no), history of falling (yes/no), and the use of walking aids will be recorded. In the evaluation of patients, Brunnstrom Hemiplegia Recovery Staging, Functional Ambulation Classification (FAC), Mini Mental State Examination(MMSE),Turkish Version of Modified Falls Efficacy Scale(MFES), Berg Balance Scale(BBS), Postural Assessment Scale for Stroke Patient Turkish Version (PASS-Turk), Modified Ashworth Scale (MAS), Modified Barthel Activities of Daily Living Index will be used. Fear of falling will be evaluated by the same researcher using the MFES. Also a question " Are you afraid of falling? (Yes/No)" will be asked. The patients will be divided into two groups as Group 1 =MFES<5 and Group2 =MFES ≥5. Balance, posture, ambulation status, spasticity, daily living activities and Brunnstrom staging will be compared between two groups. Correlation between MFES and balance, posture and activities of daily living will be studied.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 50 and over
* More than 6 months after the stroke
* Able to follow 3-digit orders
* Able to approve the consent form in writing
* Patients with a score of 23 and above on the Mini-Mental State Test will be included

Exclusion Criteria:

* Bed-dependent, wheelchair-dependent patients
* Patients diagnosed with Alzheimer's, Dementia
* Patients who are cardiovascularly unstable
* Patients with diseases that affect balance (such as Parkinson's disease, Cerebral trauma, Meniere, ear infection, Benign paroxysmal positional vertigo, Multiple sclerosis) and those who use drugs that disrupt the balance

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Chronic stroke patients, admitted to Izmir Katip Celebi University Ataturk Training and Research Hospital Physical Medicine and Rehabilitation outpatient clinic, aged 50 and older.
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2021-01-15 (Actual); Primary Completion 2022-02-01 (Actual); Study Completion 2022-02-01 (Actual)

PRIMARY OUTCOMES:
Fear of falling | 1 day (All patients will be evaluated once.)
  Fear of falling will be measured by Turkish Version of Modified Falls Efficacy Scale(MFES). It is a 14-question scale that evaluates patients' fear of falling and their self-confidence in performing daily living activities.

SECONDARY OUTCOMES:
Balance | 1 day (All patients will be evaluated once.)
  Balance will be measured by Berg Balance Scale. It consists of 14 sub-measurements. Each parameter will be evaluated by scoring between 0-4 and the total score will be revealed. Patients with a total score of 0-20 were associated with high fall risk, 21-40 moderate fall risk, 41-56 low risk
Posture | 1 day (All patients will be evaluated once.)
  Posture will be measured by Postural assessment scale for stroke patients (PASS-Turk). In the scale, there are a total of 12 parameters, 5 parameters related to maintaining posture and 7 parameters related to posture change. Each parameter will be scored between 0-3 points and the result will be the PASS-Turk Total score.
Functional Independence | 1 day (All patients will be evaluated once.)
  Functional independence will be measured by Modified Barthel Activities of Daily Living Index. It is an index that evaluates the parameters of transfer, ambulation, going up and down stairs, feeding, dressing, personal care, bathing, sitting and standing on the toilet, urine continence, stool continence and collects patients in 5 groups according to these parameter scores. In these groups evaluated between 1 and 5, 1; While it was evaluated as insufficient to do business, 5; it is evaluated completely independently.
Spasticity | 1 day (All patients will be evaluated once.)
  Spasticity will be measured by Modified Ashworth Scale. The shoulder girdle, elbow, hand, hip girdle, knee and ankle-ankle joints are scored as 0/1/1 + / 2/3/4 according to the spasticity scale by evaluating the right and left sides separately with speed-dependent passive stretching.
Hemiplegia stage | 1 day (All patients will be evaluated once.)
  Hemiplegia stage will be measured by Brunnstrom Hemiplegia Recovery Staging. This staging consists of 3 sub-headings: Upper extremity, Hand, and lower extremity. Upper extremity is evaluated from stage 1 to stage 7, hand and lower extremity from stage 1 to stage 6.
Ambulatory status | 1 day (All patients will be evaluated once.)
  Ambulatory status will be measured by Functional Ambulation Classification. Classification is evaluated between stage 0 and stage 5. Stage 5 refers to walking fully independently at any speed and on the ground.

CONTACTS AND LOCATIONS:
Overall Officials: Nese Olmez Sarikaya, Prof, Study Chair — Izmir Katip Celebi University; Bekir Tetik, MD, Principal Investigator — Izmir Katip Celebi University
Locations (1):
- Izmir Katip Celebi University, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No